CLINICAL TRIAL: NCT02339584
Title: Efficacy and Safety of Brinzolamide 10 mg/mL / Brimonidine 2 mg/mL Eye Drops, Suspension Compared to Brinzolamide 10 mg/mL Eye Drops, Suspension Plus Brimonidine 2 mg/mL Eye Drops, Solution in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy and Safety of Brinzolamide/Brimonidine Fixed Combination BID Compared to Brinzolamide BID Plus Brimonidine BID in Subjects With Open-Angle Glaucoma (OAG) or Ocular Hypertension (OHT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-13-013
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Suspensions; Ophthalmic Solutions; Solutions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brinz/Brim (Experimental): Vehicle solution, 1 drop, followed by Brinzolamide 10 mg/mL / Brimonidine 2 mg/mL fixed combination eye drops, suspension, 1 drop, administered at least 5 minutes apart in the treated eye(s) twice daily (BID) for 3 months
  Interventions: Drug: Brinzolamide 10 mg/mL / Brimonidine 2 mg/mL fixed combination eye drops, suspension; Drug: Vehicle
- Brinz+Brim (Active Comparator): Brimonidine 2 mg/mL eye drops, solution, 1 drop, followed by Brinzolamide 10 mg/mL eye drops, suspension, 1 drop, administered at least 5 minutes apart in the treated eye(s) BID for 3 months
  Interventions: Drug: Brinzolamide 10 mg/mL eye drops, suspension; Drug: Brimonidine 2 mg/mL eye drops, solution

INTERVENTIONS:
Drug: Brinzolamide 10 mg/mL / Brimonidine 2 mg/mL fixed combination eye drops, suspension
  Arms: Brinz/Brim
Drug: Brinzolamide 10 mg/mL eye drops, suspension
  Other Names: AZOPT™
  Arms: Brinz+Brim
Drug: Brimonidine 2 mg/mL eye drops, solution
  Arms: Brinz+Brim
Drug: Vehicle — Inactive ingredients used as a placebo for masking purposes
  Arms: Brinz/Brim

SUMMARY:
The purpose of this study is to compare the fixed combination (BID) [Brinzolamide 10 mg/mL / Brimonidine 2 mg/mL eyes drops, suspension] to the unfixed combination (BID) [Brinzolamide 10 mg/mL eye drops, suspension plus Brimonidine 2 mg/mL eyes drops, solution] with respect to intraocular pressure (IOP)-lowering efficacy.

DETAILED DESCRIPTION:
This study is divided into 2 phases conducted in sequence for a total of 6 visits: Phase I (Screening/Eligibility) which includes a Screening Visit, followed by 2 Eligibility Visits (E1 and E2) and Phase II (Treatment/Follow-up) which includes 3 visits at Week 2, Week 6, and Month 3. Following washout of any IOP-lowering medication, subjects who meet all inclusion/exclusion criteria at both Eligibility visits and had IOP measurements within the specified range during this period will be randomized to Phase II.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension insufficiently controlled on monotherapy or currently on multiple IOP-lowering medications;
* Mean IOP measurements within guidelines specified in the protocol. Must not be > 36 mmHg at any time point;
* Able to understand and sign an informed consent form;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, test positive for pregnancy, intend to become pregnant during the study period, breast-feeding, or not in agreement to use adequate birth control methods throughout the study;
* Severe central visual field loss in either eye;
* Unable to safely discontinue all IOP-lowering ocular medication(s) for a minimum of 5 (± 1) to 28 (± 1) days prior to E1 Visit;
* Chronic, recurrent or severe inflammatory eye disease;
* Ocular trauma within the past 6 months;
* Ocular infection or ocular inflammation within the past 3 months;
* Clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment;
* Best-corrected visual acuity (BCVA) score worse than 55 ETDRS letters (equivalent to approximately 0.60 logMAR, 20/80 Snellen, or 0.25 decimal);
* Other ocular pathology (including severe dry eye) that may preclude the administration of α-adrenergic agonist and/or topical carbonic anhydrase inhibitor (CAI);
* Intraocular surgery within the past 6 months;
* Ocular laser surgery within the past 3 months;
* Any abnormality preventing reliable applanation tonometry;
* Any conditions including severe illness which would make the Subject, in the opinion of the Investigator, unsuitable for the study;
* History of active, severe, unstable or uncontrolled cardiovascular, cerebrovascular, hepatic, or renal disease that would preclude safe administration of a topical α-adrenergic agonist or CAI;
* Recent (within 4 weeks of the E1 Visit) use of high-dose (> 1 g daily) salicylate therapy;
* Current or anticipated treatment with any psychotropic drugs that augment adrenergic response (eg, desipramine, amitriptyline);
* Concurrent use of monoamine oxidase inhibitors (MAOI);
* Concurrent use of glucocorticoids administered by any route;
* Therapy with another investigational agent within 30 days prior to the Screening Visit;
* Hypersensitivity to α-adrenergic agonist drugs, topical or oral CAIs, sulfonamide derivatives, or to any component of the study medications;
* Less than 30 days stable dosing regimen before the Screening Visit of any medications (excluding IOP-lowering treatments) or substances administered by any route and used on a chronic basis that may affect IOP, including but not limited to β-adrenergic blocking agents;
* Use of any additional topical or systemic ocular hypotensive medication during the study;
* Other protocol-specified exclusion criteria may apply.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Asia, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 26 study centers located in China (14), Russia (9), and Taiwan (3).
Pre-assignment Details: Of the 493 enrolled, 64 subjects were exited as screen failures and another 50 discontinued prior to randomization. This reporting group includes all randomized subjects (379).
Period: Overall Study
Arm/Group | Brinz/Brim | Brinz+Brim
Started | 188 | 191
Completed | 173 | 176
Not Completed | 15 | 15
Not completed — Adverse Event | 11 | 7
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received study medication, satisfied pre-randomization inclusion/exclusion criteria, and had at least 1 scheduled on-therapy study visit (Per Protocol (PP) Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinz+Brim | Total
Number analyzed (Participants) | 172 | 177 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.29) | 52.6 (16.25) | 52.4 (16.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 98 | 195
  Male | 75 | 79 | 154
Mean Diurnal Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mmHg] — IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in millimeters mercury (mmHg). Diurnal IOP was defined as the average of the three timepoints measured: 9 AM, +2 Hrs and +7Hrs. Baseline was the average of the values for 2 eligibility visits. If one of the values was missing, the other non-missing value was taken as the baseline. Only one eye (study eye) contributed to the analysis.
  mmHg | 24.62 (2.661) | 24.59 (2.660) | 24.61 (2.657)

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP Change From Baseline at Month 3
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and reported in mmHg. Diurnal IOP was defined as the average of the three timepoints measured: 9 AM, +2 Hrs and +7Hrs. Baseline was the average of the values for 2 eligibility visits. If one of the values was missing, the other non-missing value was taken as the baseline. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates greater improvement, ie, a reduction of IOP. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Month 3
Population: Per Protocol Analysis Set. Missing Month 3 data were imputed using a last observation carried forward method (LOCF).
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Brinz/Brim | Brinz+Brim
Number analyzed (Participants) | 169 | 171
mmHg | -7.2 (0.34) | -7.3 (0.34)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 134 days).
Description: An AE was defined as any untoward medical occurrence in a subject who is administered study treatment regardless of whether the event has a causal relationship with the treatment. This analysis includes all subjects who received at least 1 dose of study medication. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the protocol. Ocular AEs are presented for both study eye and non-study eye combined.
Groups:
- Brinz/Brim: All subjects exposed to Brinz/Brim
- Brinz+Brim: All subjects exposed to Brinz+Brim
Arm/Group | Brinz/Brim | Brinz+Brim
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/191
Serious Adverse Events (participants affected / at risk) | 4/188 | 4/191
Other Adverse Events (participants affected / at risk) | 12/188 | 13/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=188) | Brinz+Brim (N=191)
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=188) | Brinz+Brim (N=191)
Conjunctival hyperaemia (Eye disorders) | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.